CLINICAL TRIAL: NCT04749459
Title: Clinical Evaluation of Sunscreen Efficacy With the Sun Protection Factor Assay and Calculation of the Label SPF - ISO 24444 (2010) Test Method & Australia/New Zealand Test Method
Brief Title: Sun Protection Factor (SPF) Determination of Two Sunscreen-Containing Lip Balms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 215232
Record Dates: First submitted 2021-02-07; First posted 2021-02-11 (Actual); Results first posted 2022-03-16 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-01

CONDITIONS: Sunscreening Agents

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ChapStick Moisturizer, Classic Flavor (Experimental): This arm will include all the test sites on the participants back where ChapStick Classic Moisturizer (ANZ) will be applied.
  Interventions: Drug: ChapStick Moisturizer, Classic Flavor
- ChapStick Moisturizer, Strawberry Flavor (Experimental): This arm will include all the test sites on the participants back where ChapStick Strawberry Moisturizer (ANZ) will be applied.
  Interventions: Drug: ChapStick Moisturizer, Strawberry Flavor
- ISO 24444:2010 P2 Standard Sunscreen (Active Comparator): This arm will include all the test sites on the participants back where ISO 24444:2010 P2 Standard Sunscreen will be applied.
  Interventions: Drug: ISO 24444:2010 P2 Standard Reference Sunscreen

INTERVENTIONS:
Drug: ChapStick Moisturizer, Strawberry Flavor — A single topical application of ChapStick Moisturizer, Strawberry Flavor will be applied to the appropriate 40 square centimeter (cm^2) test site (on the back of each participants). This application shall provide a test material film of approximately 2.00 +/- 0.05 milligram per centimeter square (mg/cm^2), using 80 +/-2 milligrams (mg) of material.
  Arms: ChapStick Moisturizer, Strawberry Flavor
Drug: ChapStick Moisturizer, Classic Flavor — A single topical application of ChapStick Moisturizer, Classic Flavor will be applied to the appropriate 40 cm^2 test site (on the back of each participants). This application shall provide a test material film of approximately 2.00 +/- 0.05 mg/cm^2, using 80 +/-2 mg of material.
  Arms: ChapStick Moisturizer, Classic Flavor
Drug: ISO 24444:2010 P2 Standard Reference Sunscreen — A single topical application of ISO 24444:2010 P2 Standard Sunscreen will be applied to the appropriate 40 cm^2 test site (on the back of each participants). This application shall provide a test material film of approximately 2.00 +/- 0.05 mg/cm^2, using 80 +/-2 mg of material.
  Arms: ISO 24444:2010 P2 Standard Sunscreen

SUMMARY:
The aim of this study is to determine the SPF of two test materials ChapStick Moisturizer, Classic Flavor and ChapStick Moisturizer, Strawberry Flavor using the methodology described in the International Standard Test Method. This static methodology also meets the requirements of the Australia/New Zealand standard.

DETAILED DESCRIPTION:
A single-center, randomized, evaluator blind, intra-individual comparison, no treatment and positive controlled clinical study to determine the SPF of two ChapStick sunscreen-containing lip balms as per ISO 24444:2010. For each participant, 4 test sites will have a random assignment number for up to two test materials, control standard, and minimal erythemal dose of unprotected skin (MEDu), with at least 3 of the test sites being utilized for application. All three test sites will be exposed to UV radiation at the expected MED and subsequently evaluated for erythema 16-24 hours after UV exposure.

ELIGIBILITY:
Inclusion Criteria

* Participant must read and execute an informed consent document (that includes a HIPAA statement) indicating that the participant has been informed of all pertinent aspects of the trial before any assessment is performed;
* Participant must complete a Medical History Form (MHF) prior to their trial initiation;
* Participant must be willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other trial procedures;
* Participant must agree not to expose their back to additional sunlight or tanning beds, as either can alter the test results;
* Participant must agree not to apply any topical skin-care product to the test sites during this trial;
* Male or female participants of childbearing potential must agree to use a highly effective method of contraception throughout the trial and for 14 days after the last application of assigned treatment. A participant is of childbearing potential if, in the opinion of the investigator, he/she is biologically capable of having children and is sexually active;
* Female participants of childbearing potential must be willing to comply with urine pregnancy testing requirements prior to initiation of trial testing procedures and as may be required for the duration of the trial;
* Participant must be considered dependable and capable of understanding and following directions;
* Participant must have self-perceived Fitzpatrick skin phototype I, II, or III:

Skin Phototype Sunburn and Tanning History I Always burn easily; never tans II Always burns easily; tans minimally III Burns moderately; tans gradually; and

* Participant must have an Individual Typology Angle value >28 degrees, determined by the Testing Facility by colorimetric methods, within 1 week of trial participation.

Exclusion Criteria

* Participant is in ill health as determined by the Principal Investigator;
* Participant is an employee of the Clinical Division of the investigational site or a member of their immediate family;
* Participant is a GSK CH employee directly involved in the conduct of the trial or a member of their immediate family;
* Female participant is pregnant or intending to become pregnant over the duration of the trial or any female participant of childbearing potential who fails to produce a negative urine pregnancy test;
* Female participant who is lactating (self-reported);
* Participant using medication with photo-sensitizing potential;
* Participant has a history of adverse reactions or hypersensitivity to azo dyes, cosmetics, OTC drugs, or other topical personal care products;
* Participant taking medications other than birth control that could influence the purpose, integrity or outcome of the trial;
* Participant has used topical or systemic steroids, antihistamines, or antibiotics within 7 days of trial initiation or during the trial;
* Participant has used anti-inflammatory medications within 7 days of trial initiation or during the trial, that in the opinion of the PI, could interfere with the trial;
* Participant has used medication suspected of causing photobiological reactions (e.g., tetracyclines, thiazides, etc.), that has not been taken by the participant through a summer season;
* Participant has a dermatological condition;
* Participant has a history of abnormal response to the sun, or a condition such as lupus erythematosus or skin cancer;
* Participant uses tanning beds frequently;
* Participant whose test site was exposed to sunlight within the previous 4 weeks;
* Participant has a sunburn, suntan, uneven skin color, visible skin disease, scarring, or tattoo that would interfere with evaluation of test results; Note: The presence of non-dysplastic nevi, blemishes, or moles will be acceptable if, in the PI's judgment, they will neither compromise the clinical trial, nor jeopardize a participant's safety. A participant with dysplastic nevi should be disqualified.
* Participant has existing sun damage in the test site;
* Participant has excessive hair in the test area and are unwilling to have it clipped; or
* Participant whose test sites have been used for clinical testing in which they were exposed to ultraviolet radiation within the past 2 months.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2021-03-03 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- GSK Investigational Site, Fairfield, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months, but an extension can be granted, when justified, for up to another 12 months.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at single center in United States.
Pre-assignment Details: Total 14 participants were enrolled; up to 4 test sites on the back of each participant were randomized to treatment (2 test products, P2 Control Standard and 1 untreated site used to calculate MEDu). In total,12 participants were treated with CSM Classic (12 test sites);10 participants were treated with CSM Strawberry (10 test sites); 14 participants received P2 Control Standard (14 test sites). One participant was excluded from the final CSM Classic vs P2 Control dataset due to invalid data.
Groups:
- All Study Participants: Study participants were randomly assigned to receive a single topical application of 3 study treatments (ChapStick Moisturizer [CSM] Classic; CSM Strawberry Flavor; P2 Control Standard) or no treatment to 4 test sites on the back; 80 +/- 2 milligram (mg) product was applied to each 40 square centimeters [cm^2] test site (2.00 +/- 0.05 mg/cm^2). If there was space for only 3 test sites on the participant's back, only one of the two ChapStick products was evaluated. Test sites received a progressive sequence of timed ultraviolet radiation (UVR) exposures and were evaluated for erythema immediately after irradiation and 16-24 hours (hrs) later. A total of 14 participants were enrolled; up to 4 test sites on the back of each participant were randomized to treatment (2 test products, P2 Control Standard and 1 untreated site used to calculate MEDu). In total, 12 participants were treated with CSM Classic (12 test sites); 10 participants were treated with CSM Strawberry (10 test sites); 14 participants received P2 Control Standard (14 test sites). One participant was excluded from the final CSM Classic vs P2 Control dataset (invalid data: erythema in all sub-sites treated with the test product).
Period: Overall Study
Arm/Group | All Study Participants
Started | 14
CSM Classic | 12
CSM Strawberry Flavor | 10
P2 Control Standard | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Safety Population: all randomized participants who received at least one dose of a study treatment.
Arm/Group | All Study Participants
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Arithmetic Mean of Individual Sun Protection Factor (SPFi) Values
Description: Arithmetic mean of all valid SPFi values of each product on each participant was calculated from the individual Minimal Erythemal Dose (MED) on product treated (MEDp) test sites in relation to unprotected (MEDu) test sites 16-24 hrs after exposure to UVR. SPFi = MEDp/MEDu. No inferential statistical analysis was performed for this outcome. The MED is defined as the lowest dose of UVR that produces the first perceptible unambiguous erythema with defined borders appearing over most of the field of UVR exposure. The UVR exposure should be increased in geometric progression with 25% dose increment in relation to the expected SPF values. All individual SPF values were converted arithmetically to calculate SPF of test material (or control standard).
Time Frame: Up to 24 hours post UVR exposure
Population: All randomized participants who received study treatments (test and control standard) and provided valid SPFi values.
Measure: Mean (Standard Deviation); unit: Ratio
Groups:
- CSM Classic; P2 Control Standard (vs. CSM Classic): All participants with evaluable data for CSM Classic vs P2 Control pairwise comparison.
- CSM Strawberry Flavor; P2 Control Standard (vs. CSM Strawberry Flavor): All participants with evaluable data for CSM Strawberry Flavor vs P2 Control pairwise comparison.
Arm/Group | CSM Classic | P2 Control Standard (vs. CSM Classic) | CSM Strawberry Flavor | P2 Control Standard (vs. CSM Strawberry Flavor)
Number analyzed (Participants) | 11 | 11 | 10 | 10
Ratio | 17.3 (3.5) | 17.9 (4.4) | 19.3 (4.5) | 18.4 (4.1)
Statistical Analysis 1: Comparison: CSM Classic vs P2 Control Standard (vs. CSM Classic); Test type: Other — A minimum of 10 valid results was defined as the number required to produce mean study product (or control standard) SPF with 95% confidence interval (CI) within +/- 17% of the measured mean SPF of the study product (or control standard); CSM Classic: CIs +/- 13.7% P2 Control Standard (vs. CSM Classic) CIs +/- 16.4%
Statistical Analysis 2: Comparison: CSM Strawberry Flavor vs P2 Control Standard (vs. CSM Strawberry Flavor); Test type: Other — [test comment as in outcome 1, analysis 1]; CSM Strawberry Flavor: CIs +/- 16.6% P2 Control Standard (vs CSM Strawberry Flavour): CIs +/- 16.0%

ADVERSE EVENTS:
Time Frame: From screening until 14 days after last dose administration of trial product (Up to 29 days)
Description: Adverse events (AEs) and Serious Adverse Events (SAEs) were to be collected from time of consent until 14 days after receiving study treatment; SAEs were to be reported within 24 hrs of detection. Diagnosis was to be documented (were known), not individual signs/symptoms. AEs were to be classified by Intensity (mild, moderate, severe); Causality (probable, possible, unlikely); Serious or Non-Serious.
Arm/Group | CSM Classic | P2 Control Standard (vs. CSM Classic) | CSM Strawberry Flavor | P2 Control Standard (vs. CSM Strawberry Flavor) | All Study Participants
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/10 | 0/10 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/10 | 0/10 | 0/14
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/10 | 0/10 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-25): https://cdn.clinicaltrials.gov/large-docs/59/NCT04749459/Prot_SAP_000.pdf